CLINICAL TRIAL: NCT07389122
Title: KOBE Study: Adherence to and Tolerability of Different Very-low-calorie Ketogenic Protocols (VLCKD, Very Low-Calorie Ketogenic Diet) in Patients With Obesity and Complicated Overweight.
Brief Title: Adherence and Tolerability of Four Very Low-Calorie Ketogenic Diet Approaches in Adults With Obesity or Complicated Overweight
Acronym: KOBE
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: S. Orsola-Malpighi Hospital, University of Bologna (Unknown)
Responsible Party: Principal Investigator, Maria Letizia Petroni, Prof. Maria Letizia Petroni, University of Bologna
Other Study IDs: 650/2021/Oss/AOUBo
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); Type 2 Diabetes; Insulin Resistance
Keywords: ketogenic diet; meal replacement; pragmatic study; real-world evidence; obesity management; very-low-energy ketogenic therapy; weight loss
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2; Insulin Resistance; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm A: In arm A, protein intake was derived exclusively from natural food sources, with three or four daily meals according to individual energy and protein requirements. Protein sources included lean white meats (chicken, rabbit, turkey), lean red meats (veal and pork), lean and defatted cured meats (bresaola, cured and cooked ham), fish (gilthead seabream, cod, hake, trout), and 0% fat Greek yogurt.
- Arm B: In arm B, the same natural food sources were combined with one daily meal, corresponding to breakfast, based on whey protein supplementation.
- Arm C: In arm C, one or two daily meals, according to individual energy and protein requirements, consisted of natural foods, whereas the remaining two meals were provided as commercial meal replacement products.
- Arm D: In arm D, all daily meals consisted exclusively of commercial meal replacement products.

SUMMARY:
This study, called KOBE Study, looks at how well different very low-calorie ketogenic diets (VLCKD) are followed and tolerated by adults with obesity or complicated overweight in routine clinical practice.

Ketogenic diets are medical nutrition therapies that greatly reduce carbohydrates and calories to promote weight loss and improve metabolic health. Several VLCKD approaches are used in clinical care, but they differ in the type of protein sources used (natural foods versus meal replacements or supplements). At present, there is limited evidence comparing these approaches in terms of adherence, side effects, satisfaction, and dropout rates.

The KOBE Study is a single-center, prospective, observational study conducted during standard clinical care at a hospital nutrition clinic. Participants choose one of four VLCKD protocols based on personal preference:

* diets using only natural protein foods,
* natural proteins plus one protein supplement,
* natural proteins plus two meal replacements,
* or diets based entirely on meal replacements.

All participants follow the same structured program lasting about 26 weeks (longer for individuals with severe obesity), consisting of:

1. an initial ketogenic phase,
2. a gradual reintroduction of carbohydrates,
3. a maintenance phase based on a low-glycemic index Mediterranean-style diet. Throughout the study, patients undergo routine clinical visits and assessments, including measurements of body weight, body composition, blood tests, liver imaging, and questionnaires on hunger, bowel habits, quality of life, and satisfaction with the diet. No additional tests beyond standard care are required.

The main goal of the study is to compare the different ketogenic protocols in terms of:

* how well patients can follow them,
* how well they are tolerated,
* the occurrence of side effects,
* and overall satisfaction. Secondary objectives include evaluating changes in body composition, metabolic parameters, and liver health.

The results of this study aim to help patients and healthcare professionals make more informed, evidence-based decisions when choosing among different ketogenic diet options for weight management and metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Obesity with or without comorbidities (BMI ≥ 30 kg/m²) OR
* Overweight with comorbidity of MASLD (BMI 25.0-29.9 kg/m²) PLUS
* Previous unsuccessful attempt at a prescribed hypocaloric diet

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Breastfeeding
* Moderate or severe kidney failure
* Cardiovascular diseases: heart failure (NYHA III-IV), unstable angina, acute coronary syndrome or stroke within the past 12 months, paroxysmal atrial fibrillation, any type of atrioventricular block, left bundle branch block
* Liver diseases: Child-Pugh C, elevated transaminases with AST or ALT ≥ 5 times the upper limit of normal, INR ≥ 1.5, total bilirubin ≥ 2 mg/dL
* Diabetes: type 1 diabetes mellitus, type 2 diabetes mellitus with insufficient pancreatic endocrine reserve (C-peptide < 0.8 ng/mL), type 2 diabetes mellitus on multiple daily insulin injections
* Last attempt of VLCKD outside the research protocol within the past 12 months
* Eating disorders: anorexia nervosa, bulimia nervosa, binge eating disorder
* Psychiatric comorbidities, alcohol or substance dependence
* Frail elderly patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes all consecutive individuals who, in the context of routine clinical practice, meet the eligibility criteria for VLCKD therapy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence, collateral effects, drop-out, dietetic compliance | Until the end of the study
  The primary objective of the study is to evaluate, within routine clinical practice and by comparing four distinct VLCKD protocols, the therapeutic response of patients in terms of:
  (i) adherence (compliance), (ii) occurrence of adverse events, (iii) drop-out rate, and (iv) diet satisfaction.
  The four ketogenic protocols routinely used in patients undergoing VLCKD each consist of three phases; only the first phase differs among protocols, based on patients' personal preferences.

SECONDARY OUTCOMES:
Anthropometric Measures, Body Composition, Laboratory Parameters, and Imaging Evaluations | Until the end of the study
  The secondary objectives are to evaluate the effects of the different VLCKD protocol arms on the trends of parameters collected during routine clinical practice, including:
  (i) first- and second-level anthropometric measurements (body weight, BMI, and circumferences); (ii) body composition; (iii) biochemical laboratory tests according to the SIE Consensus Statement [8], with particular attention to serum creatinine, uric acid, and potassium levels; (iv) upper abdominal ultrasound and hepatic-splenic transient elastography assessed using the FibroScan technique.

CONTACTS AND LOCATIONS:
Locations (1):
- S.Orsola-Malpighi Hospital-University of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blake MR, Raker JM, Whelan K. Validity and reliability of the Bristol Stool Form Scale in healthy adults and patients with diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2016 Oct;44(7):693-703. doi: 10.1111/apt.13746. Epub 2016 Aug 5. PMID 27492648
- [Background] Solah VA, Meng X, Wood S, Gahler RJ, Kerr DA, James AP, Pal S, Fenton HK, Johnson SK. Effect of training on the reliability of satiety evaluation and use of trained panellists to determine the satiety effect of dietary fibre: a randomised controlled trial. PLoS One. 2015 May 15;10(5):e0126202. doi: 10.1371/journal.pone.0126202. eCollection 2015. PMID 25978321
- [Background] Gibson AA, Seimon RV, Lee CM, Ayre J, Franklin J, Markovic TP, Caterson ID, Sainsbury A. Do ketogenic diets really suppress appetite? A systematic review and meta-analysis. Obes Rev. 2015 Jan;16(1):64-76. doi: 10.1111/obr.12230. Epub 2014 Nov 17. PMID 25402637
- [Background] Caprio M, Infante M, Moriconi E, Armani A, Fabbri A, Mantovani G, Mariani S, Lubrano C, Poggiogalle E, Migliaccio S, Donini LM, Basciani S, Cignarelli A, Conte E, Ceccarini G, Bogazzi F, Cimino L, Condorelli RA, La Vignera S, Calogero AE, Gambineri A, Vignozzi L, Prodam F, Aimaretti G, Linsalata G, Buralli S, Monzani F, Aversa A, Vettor R, Santini F, Vitti P, Gnessi L, Pagotto U, Giorgino F, Colao A, Lenzi A; Cardiovascular Endocrinology Club of the Italian Society of Endocrinology. Very-low-calorie ketogenic diet (VLCKD) in the management of metabolic diseases: systematic review and consensus statement from the Italian Society of Endocrinology (SIE). J Endocrinol Invest. 2019 Nov;42(11):1365-1386. doi: 10.1007/s40618-019-01061-2. Epub 2019 May 20. PMID 31111407
- [Background] Castellana M, Conte E, Cignarelli A, Perrini S, Giustina A, Giovanella L, Giorgino F, Trimboli P. Efficacy and safety of very low calorie ketogenic diet (VLCKD) in patients with overweight and obesity: A systematic review and meta-analysis. Rev Endocr Metab Disord. 2020 Mar;21(1):5-16. doi: 10.1007/s11154-019-09514-y. PMID 31705259
- [Background] Gupta L, Khandelwal D, Kalra S, Gupta P, Dutta D, Aggarwal S. Ketogenic diet in endocrine disorders: Current perspectives. J Postgrad Med. 2017 Oct-Dec;63(4):242-251. doi: 10.4103/jpgm.JPGM_16_17. PMID 29022562
- [Background] Krebs HA. The regulation of the release of ketone bodies by the liver. Adv Enzyme Regul. 1966;4:339-54. doi: 10.1016/0065-2571(66)90027-6. No abstract available. PMID 4865971
- [Background] Westman EC, Tondt J, Maguire E, Yancy WS Jr. Implementing a low-carbohydrate, ketogenic diet to manage type 2 diabetes mellitus. Expert Rev Endocrinol Metab. 2018 Sep;13(5):263-272. doi: 10.1080/17446651.2018.1523713. PMID 30289048
- [Background] Watanabe M, Tozzi R, Risi R, Tuccinardi D, Mariani S, Basciani S, Spera G, Lubrano C, Gnessi L. Beneficial effects of the ketogenic diet on nonalcoholic fatty liver disease: A comprehensive review of the literature. Obes Rev. 2020 Aug;21(8):e13024. doi: 10.1111/obr.13024. Epub 2020 Mar 24. PMID 32207237
- [Background] Jagadish S, Payne ET, Wong-Kisiel L, Nickels KC, Eckert S, Wirrell EC. The Ketogenic and Modified Atkins Diet Therapy for Children With Refractory Epilepsy of Genetic Etiology. Pediatr Neurol. 2019 May;94:32-37. doi: 10.1016/j.pediatrneurol.2018.12.012. Epub 2018 Dec 29. PMID 30803845
- [Background] Freeman JM, Kossoff EH. Ketosis and the ketogenic diet, 2010: advances in treating epilepsy and other disorders. Adv Pediatr. 2010;57(1):315-29. doi: 10.1016/j.yapd.2010.08.003. No abstract available. PMID 21056745

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT07389122/Prot_SAP_000.pdf